CLINICAL TRIAL: NCT02914054
Title: Therapy of Adults Affected by Idiopathic Thrombocytopenic Purpura With 3 Cycles Pulses of High-dose Dexamethasone (HD-DXM)
Brief Title: Therapy of Adults Affected by Idiopathic Thrombocytopenic Purpura With Dexamethasone
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Collaborators: Adibvira (Unknown)
Responsible Party: Principal Investigator, Saeid Rezaei Jouzdani, Resident of Internal Medicine, Clinical researcher, Professional Doctor of medicine, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IUMS
Record Dates: First submitted 2016-09-19; First posted 2016-09-26 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: ITP; Croticosteroid Therapy
Keywords: ITP
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Prednisone receiving group (Active Comparator): Patients in PDN arm received PDN
  Interventions: Drug: Prednisone
- Dxamethasone receiving group (Active Comparator): In HD-DXM arm, DXM was administered
  Interventions: Drug: High dose Dexamethasone pulses

INTERVENTIONS:
Drug: High dose Dexamethasone pulses — In HD-DXM arm, DXM was administered intravenously at 40 mg in 500cc normal saline (0.9% saline) during 1 hour for consecutive 4 days and then stopped. This cycle was repeated in 14 days interval to receive 3 cycles of treatment.
  Arms: Dxamethasone receiving group
Drug: Prednisone — Patients in PDN arm received PDN orally at 1.0 mg/kg body weight daily for 4 consecutive weeks. After achieving responses the medication tapered gradually to less than 15mg daily or terminated over 4-6 weeks aimed at maintaining platelet count over 30 ×109/L.
  Arms: Conventional Prednisone receiving group

SUMMARY:
In this prospective, randomized, controlled clinical trial investigators' aim was to compare the efficacy and the adverse effect of 3 therapy cycles of HD-DXM versus conventional treatment with PDN for untreated adult patients with ITP. In this study standardized criteria and definitions were used according to consensus international working group guideline for ITPto compare clinical outcomes of the two corticosteroid treatment regimens and determine the superior regimen as a first line strategy for new primary ITP in adults

DETAILED DESCRIPTION:
Therapy of Adults affected by idiopathic thrombocytopenic purpura with 3 cycles pulses of high-dose dexamethasone (HD-DXM): a prospective randomized clinical trial Alireza Sadeghi, Saeid Rezaei Jouzdani, Forough Hosseini

Introduction :

Idiopathic thrombocytopenic purpura(ITP) is an autoimmune disorder characterized by platelet destruction leading to decreased platelet count and an increased risk of bleeding. Mechanisms including autoantibody- mediated platelet destruction, cytotoxic T-lymphocyte platelet lysis, impaired platelet maturation and production has been identified in the pathogenesis of ITP.(1)The first line treatment of ITP is still corticosteroid therapy. Prednisone(PDN) is the standard corticosteroid therapy in ITP practical guideline usually given at 1 mg/kg per day for 4 weeks and then tapered.(2) Recent studies suggested pulsed high-dose dexamethasone given at a dose 40 mg/day to a 4-day course treatment as an alternative corticosteroid instead of prednisone to reduce the duration and the adverse effect of corticosteroid therapy.(3-5) A multicenter randomized clinical trial compared the 2 corticosteroid therapy and suggested that HD-DXM has more effective and better tolerance than PDN.(4) Another multicenter cohort study using repeated courses of HD-DXM (from 6 to 4 cycles, repeated each cycle 28 days to 14 days interval) confirmed the benefit as compared with conventional therapy and proposed as a first-line treatment for patients with ITP. Also there was no difference in overall response rate between the third and the fourth cycles of HD-DXM pulses therapy, using 3 therapy cycles with 14 days interval between each cycle, has been proposed for better safety and efficacy.(5) In this prospective, randomized, controlled clinical trial investigators' aim was to compare the efficacy and the adverse effect of 3 therapy cycles of HD-DXM versus conventional treatment with PDN for untreated adult patients with ITP. In this study standardized criteria and definitions were used according to consensus international working group guideline for ITP(6) to compare clinical outcomes of the two corticosteroid treatment regimens and determine the superior regimen as a first line strategy for new primary ITP in adults.

ELIGIBILITY:
Inclusion Criteria:

* The eligible patients for this study were aged 18 or older of both genders with newly diagnosed primary ITP according to the international working group (IWG) guideline(6). All patients included in the study were treatment naïve ITP within 3 months from diagnosis and a platelet count of no more the 30×10^9/L, or more than 30×10^9/L with presence of bleeding symptoms according to the grading score of bleeding

Exclusion Criteria:

* malignancy, pregnancy or lactation, liver and kidney failure, connective tissue disorders, seropositive detection of HIV, hepatitis B virus or hepatitis C virus or any recent viral infection, active infection, diabetes, hypertension, cardiovascular disorders, autoimmune hemolytic anemia, psychosis, osteoporosis, any corticosteroid or immunosuppressive therapy in 3 months before diagnosis and any previous ITP-specific therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
platelet count | 6-12 months

CONTACTS AND LOCATIONS:
Locations (1):
- IUMS, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] McKenzie CG, Guo L, Freedman J, Semple JW. Cellular immune dysfunction in immune thrombocytopenia (ITP). Br J Haematol. 2013 Oct;163(1):10-23. doi: 10.1111/bjh.12480. Epub 2013 Aug 12. PMID 23937260
- [Background] Neunert C, Lim W, Crowther M, Cohen A, Solberg L Jr, Crowther MA; American Society of Hematology. The American Society of Hematology 2011 evidence-based practice guideline for immune thrombocytopenia. Blood. 2011 Apr 21;117(16):4190-207. doi: 10.1182/blood-2010-08-302984. Epub 2011 Feb 16. PMID 21325604
- [Background] Cheng Y, Wong RS, Soo YO, Chui CH, Lau FY, Chan NP, Wong WS, Cheng G. Initial treatment of immune thrombocytopenic purpura with high-dose dexamethasone. N Engl J Med. 2003 Aug 28;349(9):831-6. doi: 10.1056/NEJMoa030254. PMID 12944568
- [Background] Wei Y, Ji XB, Wang YW, Wang JX, Yang EQ, Wang ZC, Sang YQ, Bi ZM, Ren CA, Zhou F, Liu GQ, Peng J, Hou M. High-dose dexamethasone vs prednisone for treatment of adult immune thrombocytopenia: a prospective multicenter randomized trial. Blood. 2016 Jan 21;127(3):296-302; quiz 370. doi: 10.1182/blood-2015-07-659656. Epub 2015 Oct 19. PMID 26480931
- [Background] Mazzucconi MG, Fazi P, Bernasconi S, De Rossi G, Leone G, Gugliotta L, Vianelli N, Avvisati G, Rodeghiero F, Amendola A, Baronci C, Carbone C, Quattrin S, Fioritoni G, D'Alfonso G, Mandelli F; Gruppo Italiano Malattie EMatologiche dell'Adulto (GIMEMA) Thrombocytopenia Working Party. Therapy with high-dose dexamethasone (HD-DXM) in previously untreated patients affected by idiopathic thrombocytopenic purpura: a GIMEMA experience. Blood. 2007 Feb 15;109(4):1401-7. doi: 10.1182/blood-2005-12-015222. Epub 2006 Oct 31. PMID 17077333
- [Background] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182